CLINICAL TRIAL: NCT03681067
Title: A Phase Ib/IIb, Randomised, Double Blind, Placebo-Controlled Trial to Investigate the Safety, Tolerability and Clinical Activity of Humanised Antibody GSK1070806 in the Treatment of Patients With Moderate-to-Severe Crohn's Disease
Brief Title: A Clinical Trial of Antibody GSK1070806 in the Treatment of Patients With Moderate to Severe Crohn's Disease
Acronym: CDAID
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: GlaxoSmithKline (Industry); University Hospital Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RG_17-258; 2018-002001-65 (EudraCT Number)
Record Dates: First submitted 2018-08-20; First posted 2018-09-21 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Crohn Disease
Keywords: Crohn's disease; CDAID; CDAI; GSK1070806
MeSH Terms: conditions — Crohn Disease | interventions — GSK1070806

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GSK10708060 (Experimental): Humanised antibody GSK1070806
  Interventions: Drug: GSK1070806
- Placebo - sodium chloride (Placebo Comparator): Placebo
  Interventions: Drug: Placebo- sodium chloride

INTERVENTIONS:
Drug: GSK1070806 — GSK1070806 100mg/ml injectable solution will be delivered via intravenous infusion as a single infusion
  Arms: GSK10708060
Drug: Placebo- sodium chloride — Placebo injectable solution will be delivered via intravenous infusion as a single infusion
  Other Names: Placebo
  Arms: Placebo - sodium chloride

SUMMARY:
This trial aims to investigate the safety, tolerability and clinical activity of humanised antibody GSK1070806 delivered via intravenous infusion in the treatment of patients with moderate-to-severe Crohn's disease. 30-36 patients will be enrolled into the trial, with two thirds of the patients receiving active drug and one third receiving placebo. After 30 patients have been recruited into the study the sample size will be reassessed and up to an additional 6 patients could be recruited (i.e. up to 36 patients).

DETAILED DESCRIPTION:
The proposed study will be a randomised, double blind, placebo-controlled trial to investigate the safety, tolerability, clinical activity, pharmacokinetics and pharmacodynamics of single intravenous infusion (one dose on Day 1) of GSK1070806 or placebo, in patients with active, moderate to severe CD. The primary objective of the study is to assess the safety and tolerability of a single dose IV administration of GSK1070806. A secondary objective will be to evaluate the effect of GSK1070806 in change of CDAI over time. Further secondary endpoints will include assessment of endoscopic response in patients at week 12. (Other secondary endpoints are detailed in Section 2.3).

30 patients will be recruited with randomisation of 2:1 active drug to placebo in multiple centres in the UK. After 30 patients have been recruited into the study the sample size will be reassessed and up to an additional 6 patients could be recruited (i.e. up to 36 patients). These additional patients will also be recruited with randomisation of 2:1 active drug to placebo.

An initial screening shall take place to identify patients diagnosed with CD for at least 3 months prior to screening, active disease based on CDAI score of 220-450 points and colonoscopic confirmation of active mucosal inflammation (SES-CD excluding narrowed component ≥6; or in patients with isolated ileal disease ≥4).

Patients who do not have colonoscopically demonstrated mucosal inflammation will be excluded even if they have MRI evidence of Crohn's disease more proximally in the small intestine. For inclusion, CDAI criteria have to be fulfilled within 7 days prior to dosing and colonoscopic SES-CD criteria has to be fulfilled with 28 days prior to dosing.

The induction of clinical activity will be assessed at week 12 by CDAI score, average clinical SF and/or AP scores as well as by colonoscopic assessment of baseline video images and week 12 video images.

The first 5 patients randomised into the trial will be dosed at least 3 days apart. At the interim analysis time point, a safety decision will be taken on the subsequent recruitment and patient spacing out strategy.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for inclusion in this study only if all of the following criteria apply:

1. Written informed consent prior to any of the screening procedures including discontinuation of prohibited medications. (see Section 7.11 for additional information)
2. Patients that have been diagnosed with moderate to severe Crohn's disease for at least 3 months prior to Screening Visit 1
3. Patients are required to have endoscopic evidence of active Crohn's disease at Baseline defined by endoscopic appearance: SES-CD excluding the narrowed component of ≥ 6 (or ≥4 for patients with isolated ileal disease).
4. AST and ALT ≤ 2xULN; alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
5. Male or female participants aged ≥16 years (up to 80 years)

   Male participants:
6. A male participant must agree to use contraception as detailed in Appendix 5 of this protocol for at least 180 days post-dose of study medication and refrain from donating sperm during this period.

   Female participants:
7. If the patient is breastfeeding, she must agree to stop breastfeeding once randomised into the trial.*
8. A patient is eligible to participate if she is not pregnant.
9. A woman of childbearing potential (WOCBP) is eligible only if she meets at least one of the following conditions:

   i. Females on HRT and whose menopausal status is in doubt will be required to use one of the non-hormonal highly effective contraception methods if they wish to continue their HRT during the trial. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before trial enrolment.

   ii. Agrees to follow the contraceptive guidance in Appendix 5 for at least 180 days post-dose of trial medication. If a hormonal method of birth control is selected from the list in Appendix 5 then patients must have been using these methods at least 1 month prior to GSK1070806 administration, or be abstinent, or utilise a condom as a method of contraception until the selected hormonal method has been in place for the 28 day period.
10. A woman who is not of childbearing potential is eligible only if she meets at least one of the following conditions:

    i. Premenopausal female with documented hysterectomy ii Premenopausal female with documented bilateral salpingectomy or oophorectomy iii. Postmenopausal female defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement

    * A female patient who is breastfeeding may be screened. If randomised into the trial, this patient must agree to stop breastfeeding. Patients who are screened but ineligible can continue breastfeeding.

therapy (HRT). However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

Exclusion Criteria:

A participant will not be eligible for inclusion in this trial if any of the following criteria apply:

1. Diagnosis of ulcerative or indeterminate colitis

   Crohn's Disease complications:
2. Evidence of an infected abscess by MRI or other examinations
3. Bowel surgery other than appendectomy within 12 weeks prior to screen and/or has planned surgery or deemed likely to need surgery for CD during the trial period
4. Participants with ileostomies, colostomies or rectal pouches
5. Participants with a bowel stricture that is fixed
6. Participants with evidence of short bowel syndrome
7. Participants requiring enteral or parenteral feeding
8. Deep penetrating ulcers at endoscopy thought to be at risk for perforation

   Viral and bacterial infections:
9. Presence of Hepatitis B surface antigen (HBsAg), (confirmed by Hepatitis B surface antigen test - within 12 months of randomisation) core antigen (HBcAg) or surface antibody (HBsAb), positive Hepatitis C (qualitative enzyme immunoassay) test result
10. Known varicella, herpes zoster, or other severe viral infection within 6 weeks of randomisation
11. The participant has a history of tuberculosis (TB) disease or latent TB infection, in the absence of documented adequate therapy for same.
12. Positive screening test for TB (including T-SPOT.TB TB test), unless respiratory review confirms false positive test results
13. History of uncontrolled bacterial or fungal infection requiring intravenous antibiotics
14. Positive immunoassay for Clostridium difficile toxin and other enteric pathogens

    Other exclusion criteria:
15. Cardiology assessment/co-morbidity defined as:

    i. QTc >450 msec (480msec for those with Bundle Branch Block) and/or ii. either QTcb or QTcf, machine or manual overread, males or females. The QT correction formula used to determine exclusion and discontinuation should be the same throughout the trial and/or iii. based on single QTc value (average of triplicate readings) of ECG obtained over a brief recording period
16. The participant has congenital or acquired immunodeficiency, or a history of chronic or recurrent opportunistic infections
17. The participant has current evidence of, or has been treated for a malignancy within the past five years (other than localised basal cell, squamous cell skin cancer, cervical dysplasia, or cancer in situ that has been resected)
18. Use of any investigational drug within 30 days prior to screening, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
19. Participant has received live, attenuated or recombinant vaccine(s) within 2 months of randomisation or will require vaccination within 3 months of trial drug infusion
20. Any patients that are receiving medication(s) detailed in Section 7.11.2 of the trial protocol, will not be eligible for randomisation into the trial

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability parameters include: adverse events and serious adverse events | 24 weeks
  NCI-CTCAE criterion Version 4
Safety and tolerability parameters include: clinical laboratory tests (Haematology) | 24 weeks
  Haematology panel : haemoglobin (g/L), Platelets (10*9/L), White Blood Cells (10*9/L), International normalized ratio, Neutrophils (10*9/L)
Safety and tolerability parameters include: clinical laboratory tests (Biochemistry) | 24 weeks
  Biochemistry Panel : Creatinine (umol/L), Sodium (mmol/L), Potassium (mmol/l), Bilirubin (umol/L), Alanine Transferase (u/L) Aspartate Transaminase (U/L), Albumin (g/L), eGFR ml/min/1.7, C-Reactive Protein (CRP)
Safety and tolerability parameters include: Cardiology | 24 weeks
  Electrocardiogram review - for any abnormalities i.e. QT interval etc.
Safety and tolerability parameters include: frequency, type and severity of infections | 24 weeks
  NCI-CTCAE criterion Version 4 - grading system used
Safety and tolerability parameters include: Heart Rate (vital signs) | 24 weeks
  Heart rate
Safety and tolerability parameters include: Blood Pressure (vital signs) | 24 weeks
  Blood pressure
Safety and tolerability parameters include: Body Temperature (vital signs) | 24 weeks
  Oral body temperature
Safety and tolerability parameters include: Respiratory Rate (vital signs) | 24 weeks
  Respiratory rate

SECONDARY OUTCOMES:
CDAI score over time. Patients | 28 weeks
  Crohns disease activity index score (Pre-treatment, Post treatment). Scale ranges from <150(remission) to >450(severe Crohn's disease).

CONTACTS AND LOCATIONS:
Overall Officials: Marietta Iacucci, MD,PhD, Principal Investigator — University of Birmingham
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, United Kingdom